CLINICAL TRIAL: NCT04430972
Title: Is Pre-operative Impaired imMune rEsponsiveness Associated With Adverse Outcome Following Aortic Valve Replacement SURgEry (MEASURE)
Brief Title: Immune Responsiveness and Outcome After Aortic Valve Surgery (Measure)
Acronym: Measure
Status: Not yet recruiting | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 263703
Record Dates: First submitted 2020-05-20; First posted 2020-06-16 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Aortic Valve Disease; Surgery--Complications; Immune System Disorder
Keywords: staphylococcus; EndoCAb; Immunity; Cardiac Surgical Procedure; sepsis
MeSH Terms: conditions — Aortic Valve Disease; Immune System Diseases; Sepsis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum Plasma PaxGene for genetic sequencing Monocytes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Aortic valve replacement — Open surgical replacement of aortic valve

SUMMARY:
There is considerable morbidity and mortality associated with cardiac surgery. Currently little effort is made to quantify how well the immune system of an individual can cope with inflammation or infection to which they are exposed during surgery.

The investigators have previously demonstrated that having higher pre-operative antibody levels is associated with a lower risk of infection and a shorter stay in hospital after cardiac surgery.

The investigators aim to study 150 patients undergoing aortic valve replacement and explore their dynamic immune responsiveness. The investigators will determine if this response is correlated with the post-operative outcome (development of post-operative infection or increased length of hospital stay).

The investigators will compare this response with the previously measured static markers of immune competence and also with a novel device that may give a more rapid measure of dynamic immunity.

The investigators will approach patients in the cardiac surgical pre-assessment clinic to see if they are willing to participate in the study.

Immediately once under anaesthetic blood will be taken for testing and then again at the end of surgery, 24h after surgery, at discharge from hospital, and at follow-up clinic approximately 4 weeks later. There will be no additional needle insertions on top of those routinely performed. The investigators will collect data from the routine observations as far as 1 year after surgery.

If the investigators can show an association between immune function and subsequent post-operative outcome it may be possible to determine ways to improve outcomes for patients undergoing heart surgery.

This might include better information on risks and benefits of surgery, actively boosting immune function (vaccination, immune-nutrition), passively improving immunity (administering antibodies), or consider current alternatives to open heart surgery where the threat of infection or inflammation may be markedly reduced (eg trans-catheter aortic valve implantation)

DETAILED DESCRIPTION:
Experimental design and methods:

Setting:

Barts Heart Centre is a 255-bedded specialist cardiac centre where approximately 200 primary isolated open aortic valve replacement procedures are performed per year. It is closely associated both geographically and academically with the William Harvey Research Institute (WHRI), which forms part of Queen Mary University, London (QMUL). This will allow laboratory analysis of all collected blood samples within 15 minutes if necessary. Barts Heart Centre is one of the largest cardiac units in Europe and a key research objective of QMUL/WHRI is to support cardiac research.

Sample collection and storage:

Following written informed consent all patients will be pre-operatively risk-scored by means of ASA, Euroscore 2 and conventionally risk-scored for the development of surgical site infection.

Blood (44ml total) will be taken from 150 aortic valve replacement patients immediately prior to surgery (T0).

Blood (7ml) will be collected into a PAXgene tube and stored at -80° for later genetic analysis. A clotted sample (7ml) will be collected in a standard gold top SST tube, left to clot then centrifuged for 10 mins at 1000g, the serum separated and stored at -80° for later analysis of antibody levels. In addition, 30 ml blood will be taken for study of peripheral blood mononuclear cells (PBMCs), drawn into standard purple top EDTA tubes (anticoagulant). These will be separated within 3 hours of collection by Ficoll-Paque density gradient centrifugation, whereby PBS-diluted blood is carefully layered over Ficoll and spun brake off in a centrifuge at 400g for 30 minutes. The PBMC layer is then extracted and washed twice in PBS and stored in 10% dimethyl sulfoxide freezing solution in liquid nitrogen so that they can be thawed, and batch analysed at a later date.

Sample analysis:

PBMCs will be counted using a haemocytometer, then cultured in RPMI and 10% serum with either LPS, α-toxin or unstimulated for 24 hours, after which they will be analysed immediately as detailed below.

• Soluble Mediators (Plasma)

* Storage: Ethylenediaminetetraacetic acid (EDTA, BD Biosciences Vacutainer, 9mL) anticoagulated blood will be centrifuged (1200g, 10mins, 20°C) and plasma stored at -80°C within 2hrs of collection
* Analysis:

Cytokines: Meso Scale Discovery (MSD) V-PLEX Proinflammatory Panel 1 will be employed to quantify IFN-γ, IL-10, IL-12p70, IL-13, IL-1β, IL-2, IL-4, IL-6, IL-8, and TNF-α. Plates will be read using a MSD QuickPlex SQ 120 imager (Wiliam Harvey Institute, QMUL).

Antibodies: These will be measured by means of ELISA assays against staphylococcal antigens (α-toxin, teichoic acid) and core moieties of the endotoxin molecule (EndoCAb).

* Whole blood LPS/α-toxin Stimulated Cytokine Release

  * Technique: As previously described and validated in our laboratory, heparinized blood will be stimulated for 4hrs (37°C, 250rpm) with 1ng/ml LPS within 2hrs of draw. After incubation, samples will be centrifuged (1200g, 10mins, 20°C) and supernatant stored at -80°C.
  * Cytokine quantification: As per 'soluble mediators' MSD V-PLEX Proinflammatory Panel 1 will be employed to quantify TNF-α (primary outcome as metric of immune competence) and other cytokines. Cytokines will be expressed as a factor of the number of circulating monocytes.
* Flow Cytometric Immunophenotyping and Functional Assessment of Leukocytes

  * Flow Cytometry: All samples will be analysed on the same machine (Becton Dickinson (BD) Fortessa, Rayne Building, UCL). Standardisation and comparison of output will be achieved via employment of constant voltages and compensation matrix throughout with daily matching of values to a single batch of Cytometry Setup and Tracking (CS&T) beads (BD). Leukocyte cell surface staining will be conducted using antibodies principally supplied by BD. Staining, data capture and storage will be conducted in accordance with a single study standard operating procedure. 5 panels (up to 14-colour) and two functional assays will be performed at each time-point. Data will be analysed in FlowJo version 10.5.
  * Surface Marker Staining:

Quantification and calibration panel: CD45, CD56, CD3, CD4, CD8, CD19, CD14, CD16, performed in a BD TruCount tube to enable enumeration of cell subsets Cell specific panels (incorporating markers of sub-categorisation and markers of immune competence)

* Monocyte/Myeloid: CD3, CD19, CD56, CD163, CD16, CD33, CD141, CD206, CD274, CD14, CD1c, CD11c, HLA-DR, CD80, CD123, CD83
* Neutrophil: CD3, CD19, CD56, HLA-DR, CD64, CD62L, CD11b, CD88, CD66b, CD14, CD11c, CD16, CD184, CD182
* Lymphocyte: CD19, CCR6, CD45RA, CD3, CD4, CD8, CXCR3, CD127, CD62L, CD25, CD56, CD27, CD279 HLA-DR Expression: Will be quantified on CD14+ monocytes using BD QuantiBrite beads.

  * Functional Measures Phagocytosis: The ability of neutrophils and monocytes to phagocytose opsonised FITC-labelled E.coli bacteria will be quantified via the PhagoTest assay (BD) as per manufacturer's instructions Reactive oxygen 'burst': Quantitative determination of leukocyte oxidative burst will be undertaken using the PhagoBurst assay (BD) in response to un-labelled opsonized E.coli, phorbol 12-myristate 13-acetate (PMA) and the chemotactic peptide N-formyl-Met-Leu-Phe (fMLP).

o The pre-surgery sample PBMCs that will be stimulated with LPS (type and concentration to be optimized via dose response curve on healthy volunteers) and α-toxin will undergo flow cytometry to measure TLR4 and TLR5 surface expression, HLA-DR surface expression and quantification of NF-kB using appropriate antibodies validated in the literature. At the end of stimulation, cells will be harvested, and RNA extracted for quantitative (q)PCR to evaluate AID mRNA expression. Although B cells in the PBMC cultures have been stimulated in the presence of other cell types, primarily T cells and monocytes-macrophages, our endpoint is to measure a B-cell response, as AID is exclusively expressed in B cells.

Enough healthy volunteer blood is available so that all above techniques can be adequately practiced and optimized prior to patient recruitment.

Further sampling timepoints will be immediately post-op (T1), 24h post-op (T2), discharge (T3) and 4 weeks post-op at surgical follow up (T4). The blood collected at 4-week post-surgery follow up will be assayed for IgG antibody assay to EndoCAb, α-toxin and teichoic acid. This will enable a measure of class switch recombination. Which will be referable back to the degree of expression of AID mRNA.

The population of aortic valve replacement patients will be followed up for mortality and major morbidity. They will be scored as per C-POMS (cardiac post-operative morbidity score), length of ITU stay and length of hospital stay. Patients will be monitored for development of surgical site infection (SSI) or the acquisition of post-operative hospital acquired infection (HAI). Post-discharge follow-up for wound infection or breakdown will be continued for 12 months.

At the immediately pre-operative timepoint (T0), alongside currently accepted measures of immune responsiveness it is intended to perform a near patient test of immune responsiveness (LIT) using a handheld chemiluminescence device that relies upon leukocyte oxidative burst to a supramaximal stimulus (Oxford Medistress). This relies upon analysis of the response in a 10mcl fresh capillary blood sample.

Statistical considerations:

From published data from centres worldwide it is known that a proportion of patients develop an infection, either surgical site infection (SSI) or hospital acquired infection (HAI), following aortic valve surgery. It is also known that these patients endure longer stay in hospital following surgery.

The investigators have demonstrated that amongst these patients there is variability in levels of antibodies to various perioperative threats, namely endotoxin and staphylococcus.

The investigators have demonstrated that in the patients who are undergoing surgery and have low levels of circulating antibody to endotoxin and/or staphylococcus there is an association with greater likelihood of developing an infection and a longer length of post-operative stay. The investigators estimate that the rate of infection varies between 13.5 - 33%.

The investigators have previously suggested that the association between antibody level and outcome may be manifestation of an underlying impaired ability in some individuals to mount a normal immune response to these threats.

It is known that a proportion of individuals have an abnormal immune response. This is perhaps most obviously seen in the response to vaccination where previous work has demonstrated the lack of immune responsiveness following various vaccination programs and our own work on EndoCAb response to monovalent typhoid vaccination. This non/poor responsiveness in these studies lies somewhere between 10 and 40%. The diagram illustrates the proportion of non-responders (ie poor immune responsiveness) if they are equally distributed.

ELIGIBILITY:
Inclusion Criteria:

• Patients undergoing first-time open aortic valve replacement surgery

Exclusion Criteria:

* Age less than 18y (capacity to consent)
* Ongoing sepsis (immunomodulatory effects, established influence on outcome from surgery)
* Immunosuppressive therapy
* Suffering from known immunosuppressive disease
* Pregnancy (immunosuppressive aspects to pregnancy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients undergoing first-time aortic valve replacement that do not fulfil any of the exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants who develop any post operative, healthcare associated infection. | Development of a HealthCare Associated Infection (HCAI) will be evaluated at one year from date of discharge from hospital.
  Development of post-operative healthcare associated infection as defined in the Centre for Disease Control and National Healthcare Safety Network guidance.

SECONDARY OUTCOMES:
Post-operative length of stay | Will be assessed at study completion, at one year following discharge from hospital.
  Time spent in hospital following surgery measured in days
Correlation of pre-operative antibody levels with in vitro immune response profiles | 2 years
  Determining if there is a correlation between those patients with low antibody levels pre-operatively to endotoxin core and staphylococcal epitopes with the dynamic immune responsiveness in an in vitro test of immune response
Does the result from a simple, point of care test of immune function correlate with that from a more comprehensive, laboratory based test of immune function | 2 years
  To determine whether the result obtained from a bedside test of immune function (LITTM) correlates with the result obtained from an in-vitro, laboratory-based test of immune function.
  The bedside test relies on the chemiluminescence result from a supramaximal stimulus of neutrophils and gives a result in the form of a continuous variable, allowing the ranking of the subjects in order of their neutrophil responsiveness.
  The laboratory-based tests, performed using flow cytometry, will look at the immune function of monocytes and each assay of a number of cytokines and cell markers will give results as a continuous variable. This again will allow for an overall ranking of patients in terms of the value obtained for each parameter measured. Participants will also be ranked according to the summed rank positions for each variable.
  Correlation between the rank order of patients determined by the two separate assays of function will be compared by calculating correlation coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Thiemermann, Study Director — Queen Mary University London
Locations (1):
- St Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Smith A, Moravcova S, Treibel TA, Colque-Navarro P, Mollby R, Moon JC, Hamilton-Davies C. Relationship between endotoxin core, staphylococcal and varicella antibody levels and outcome following aortic valve replacement surgery: a prospective observational study. Perioper Med (Lond). 2018 Sep 20;7:20. doi: 10.1186/s13741-018-0101-z. eCollection 2018. PMID 30250733
- [Result] Moravcova S, Kyle B, Shanahan H, Giannaris S, Smith A, Hamilton-Davies C. Variability of anti-staphylococcal antibodies in healthy volunteers and pre-cardiac surgery patients. Perioper Med (Lond). 2016 May 27;5:13. doi: 10.1186/s13741-016-0039-y. eCollection 2016. PMID 27239299
- [Result] Hamilton-Davies C, Barclay GR, Cardigan RA, McDonald SJ, Purdy G, Machin SJ, Webb AR. Relationship between preoperative endotoxin immune status, gut perfusion, and outcome from cardiac valve replacement surgery. Chest. 1997 Nov 5;112(5):1189-96. doi: 10.1378/chest.112.5.1189. PMID 9367456
- [Result] Bennett-Guerrero E, Ayuso L, Hamilton-Davies C, White WD, Barclay GR, Smith PK, King SA, Muhlbaier LH, Newman MF, Mythen MG. Relationship of preoperative antiendotoxin core antibodies and adverse outcomes following cardiac surgery. JAMA. 1997 Feb 26;277(8):646-50. PMID 9039883
- [Result] Hamilton-Davies C, Barclay GR, Murphy WG, Machin SJ, Webb AR. Passive immunisation with IgG endotoxin core antibody hyperimmune fresh frozen plasma. Vox Sang. 1996;71(3):165-9. doi: 10.1046/j.1423-0410.1996.7130165.x. PMID 8912459
- [Result] Poland GA, Ovsyannikova IG, Jacobson RM. Vaccine immunogenetics: bedside to bench to population. Vaccine. 2008 Nov 18;26(49):6183-8. doi: 10.1016/j.vaccine.2008.06.057. Epub 2008 Jul 1. PMID 18598732